CLINICAL TRIAL: NCT07095218
Title: Modulation of Cross-Frequency Theta-Gamma Coupling Via Gamma Transcranial Alternating Current Stimulation in Healthy Adults
Brief Title: Gamma Transcranial Alternating Current Stimulation in Healthy Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, FATMA AYDIN, Msc, Medipol University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: E-10840098-202.3.02-2205
Record Dates: First submitted 2025-07-07; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Healhty
Keywords: gamma; tACS; theta-gamma coupling

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 80 Hz Group (Experimental): transcranial alternating current stimulation (tACS) at 80 Hz gamma frequency will be applied to the bilateral dorsolateral prefrontal cortex (DLPFC) in a single 20-minute session.
  Interventions: Device: Application of Tacs
- 40 Hz Group (Experimental): transcranial alternating current stimulation (tACS) at 40 Hz gamma frequency will be applied to the bilateral dorsolateral prefrontal cortex (DLPFC) in a single 20-minute session.
  Interventions: Device: Application of Tacs
- Individual gamma Group (Experimental): transcranial alternating current stimulation (tACS) at ındividual (Hz) gamma frequency will be applied to the bilateral dorsolateral prefrontal cortex (DLPFC) in a single 20-minute session.
  Interventions: Device: Application of Tacs
- 6-80 Hz Group (Experimental): transcranial alternating current stimulation (tACS) at 6-80 Hz will be applied to the bilateral dorsolateral prefrontal cortex (DLPFC) in a single 20-minute session.
  Interventions: Device: Application of Tacs
- Sham Group (Placebo Comparator): transcranial alternating current stimulation (tACS) at sham will be applied to the bilateral dorsolateral prefrontal cortex (DLPFC) in a single 20-minute session.
  Interventions: Device: Application of Tacs

INTERVENTIONS:
Device: Application of Tacs — In this study, a single 20-minute session of tACS will be administered over the bilateral dorsolateral prefrontal cortex (DLPFC) at various gamma frequencies (40 Hz, 80 Hz, individual gamma frequency) and in a theta-gamma coupling range (6-80 Hz). A sham stimulation group will also be included. The anodal surface electrode will be placed over the left DLPFC (F3 according to the 10-20 system), and the cathodal electrode over the right DLPFC (F4). Pre- and post-stimulation cognitive performance will be assessed using neuropsychological tests, while EEG will be used to evaluate theta-gamma phase-amplitude coupling and oscillatory changes.

SUMMARY:
Transcranial Alternating Current Stimulation (tACS), particularly at gamma frequencies, may enhance fast brain oscillations (especially gamma and possibly beta), while reducing slower rhythms such as theta. These effects are not confined to the stimulation site (e.g., the precuneus) but can extend to structurally and functionally connected regions, including the default mode network (DMN). Notably, 40 Hz gamma tACS applied to the left dorsolateral prefrontal cortex (DLPFC) has been associated with improvements in working memory and motor learning during reaction time tasks. While beta-frequency stimulation often shows no significant effect, gamma-frequency tACS has been shown to reduce response times.

Gamma oscillations are commonly disrupted in neuropsychiatric disorders. These rhythms depend on a balance between excitation and inhibition, possibly linked to interneuron dysfunction. Abnormal gamma activity has been proposed as a biomarker for cognitive impairment. In this context, non-invasive rhythmic stimulation aiming to restore gamma activity is a promising cognitive enhancement strategy, though unlike pharmacological approaches, gamma-tACS has not yet been widely adopted in clinical practice.

A meta-analysis of 56 studies emphasized that tACS outcomes vary with stimulation frequency, brain region, and timing protocols. Research suggests that the susceptibility of gamma oscillations to external modulation may provide insights into cognitive reserve, domain-specific processes, and Alzheimer's disease progression. Oscillatory changes may help predict conversion from MCI to Alzheimer's disease. However, evidence on the neural mechanisms of tACS remains limited and heterogeneous, and outcomes appear to depend on task type, frequency, and intensity.

In this study, we will deliver a single 20-minute tACS session over the bilateral DLPFC using gamma frequencies (40 Hz, 80 Hz, and individualized gamma), and a theta-gamma coupling range (6-80 Hz). A sham group will also be included. The anodal electrode will be placed over F3, and the cathodal electrode over F4 (10-20 system). Cognitive performance will be assessed pre- and post-stimulation using neuropsychological tests, and EEG will measure theta-gamma phase-amplitude coupling and changes in oscillatory activity.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 40 years of age
* Scoring above 25 on the Montreal Cognitive Assessment (MoCA)
* Being right-handed
* Having no history of neurological or psychiatric diagnosis

Exclusion Criteria:

Having a neurological or psychiatric disorder

Use of medications with sedative or stimulant effects

Presence of metal brain implants or a pacemaker

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Öktem Verbal Memory Test | Before and immediately after applying Tacs
  Öktem Verbal Memory Test is a test of verbal memory processes, developed and validated by Öktem in 1992. It is designed to measure various variables related to memory.
Resting State EEG and TASK EEG | Before and immediately after applying Tacs
  The EEG recordings of the participants will be conducted using a BrainAmp 64-channel DC system. A 64-channel EasyCap will be used. AFz will serve as the ground electrode, and FCz will be used as the reference electrode. Impedance values will be maintained below 10 kOhm. EEG data will be recorded using the BrainVision Recorder software (Brain Products, Munich, Germany) with a band-pass filter set between 0.01 and 250 Hz.A 4-minute eyes-open and a 4-minute eyes-closed resting-state EEG recording will be conducted. EEG will also be recorded during the 2-back task and the memory task.
  2-back Task: A visual n-back task will be administered to assess working memory. The task load will consist of 8-minute sessions.
  Memory Task:
  The memory task, which involves both encoding and retrieval of episodic information, will be examined using a visual memory paradigm presented to the participants.
Forward and Backward Digit Span | Before and immediately after applying Tacs
  This test, which is a subtest of the Wechsler Memory Scale, was developed to assess overall attention. It consists of two stages. The first stage evaluates the forward digit span, composed of random sequences ranging from 2 to 8 digits. In the second stage, the backward digit span is assessed using random sequences of 2 to 7 digits. In the first stage, numbers are read aloud with one-second intervals, and participants are expected to repeat the sequences exactly as presented. In the second stage, numbers are again read with one-second intervals, but participants are required to repeat the digits in reverse order. The test is terminated if the participant makes consecutive errors. The forward digit span assesses sustained attention, while the backward span also evaluates working memory performance.
Verbal fluency tests | Before and immediately after applying Tacs
  Verbal fluency tests measure the ability to generate words within a specific category over a limited time period. Verbal fluency performance has been associated not only with general language skills and semantic memory functions but also with executive functions such as attention, working memory, and processing speed. In this study, semantic and phonemic fluency tasks will be used.

OTHER OUTCOMES:
Montreal Cognitive Assessment (MoCA) | Just before joining the study
  The Montreal Cognitive Assessment (MoCA) is a widely used tool designed to evaluate individuals' cognitive functions. The test scores range from a minimum of 0 to a maximum of 30. In the MoCA, higher scores indicate better cognitive performance, while lower scores may suggest the presence of cognitive impairment. In clinical practice, a score of 26 or above is generally considered indicative of normal cognitive functioning, whereas scores below 26 may reflect mild cognitive impairment. Additionally, it is recommended to add 1 point to the total score for individuals with 12 years of education or less. Scores between 18-25 are typically associated with mild cognitive impairment, scores between 10-17 with moderate impairment, and scores between 0-9 with severe cognitive impairment. However, MoCA test results should always be interpreted in conjunction with comprehensive clinical evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Lütfü Hanoğlu, Study Director — Medipol University
Locations (1):
- Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided